CLINICAL TRIAL: NCT01844947
Title: An Exploratory Phase I Study With Sorafenib in Addition to Vinflunine in Progressive Locally Advanced or Metastatic Transitional Cell Carcinoma of the Urothelial Tract
Brief Title: Phase I Study With Sorafenib in Addition to Vinflunine in Metastatic Transitional Cell Carcinoma of the Urothelial Tract
Acronym: VINSOR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr Anders Ullén (Other)
Collaborators: Bayer (Industry); Pierre Fabre Laboratories (Industry); Nordic Urothelial Cancer Oncology Group (Unknown)
Responsible Party: Sponsor-Investigator, Dr Anders Ullén, Associate Professor/Sr Consultant Clinical Oncology, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NUCOG III; 2011-004289-14 (EudraCT Number)
Record Dates: First submitted 2012-11-05; First posted 2013-05-03 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Urothelial Carcinoma; Bladder Cancer; Renal Pelvis Cancer; Ureter Cancer; Urethra Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — vinflunine; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vinflunine + sorafenib (Experimental): Single arm study.
  Interventions: Drug: Vinflunine; Drug: Sorafenib

INTERVENTIONS:
Drug: Vinflunine — Vinflunine (Javlor®, Pierre Fabre Pharma): 320 mg/m2 I.V., day 1, repeated every 21 days for patients with PS 0, adequate renal (creatinine clearance >60 ml/min) and hepatic function (as described in the inclusion criteria). PLEASE NOTE THAT THE 320 mg/m2 ARM IS CLOSED FOR RECRUITMENT.
  For patients with PS 1, or age 75 to 80 years, or exposed to radiation of the lower pelvis region, or with impaired renal function (creatinine clearance 40-60 ml/min) but adequate hepatic function (as described in the inclusion criteria), the dose of vinflunine is 280 mg/m2 I.V. day 1, repeated every 21 days.
  Other Names: Javlor
Drug: Sorafenib — Sorafenib (Nexavar®, Bayer HealthCare) daily dosage from day 2 through day 21 (repeated every 21 days):
  Step 1: 400 mg P.O. (i.e. one (1) tablet 200 mg morning and evening, 1+0+1) Step 2: 600 P.O. (i.e. one (1) tablet 200 mg morning and two tablets evening, 1+0+2) Step 3: 800 mg P.O. (i.e. two (2) tablets 200 mg morning and evening, 2+0+2) Doses of sorafenib higher than 400 mg P.O. b.i.d. are not allowed.
  Other Names: Nexavar

SUMMARY:
This study aims to analyse the tolerability (side effects and safety) with standard treatment (Javlor®) with the addition of a second anti-tumour drug: sorafenib (Nexavar®). This is the first time this treatment combination is studied in humans. Samples of blood, urine and tumour tissues will be analysed for molecular biomarkers. These biomarkers may potentially help us in the future in predicting whether a patient will benefit or not from the cancer treatment. The study also aims to investigate if a newer imaging method, called PET-CT (positron emission tomography-computed tomography), at an earlier stage (than a normal CT scan) can identify patients who will benefit from the given treatment.

DETAILED DESCRIPTION:
Objectives

* To explore the safety of sorafenib in combination with vinflunine in patients with transitional cell carcinoma of the urothelial tract and to define a recommended phase II dose for this treatment combination
* To correlate early tracer 18F-FDG-PET/CT functional imaging readouts with standard RECIST (version 1.1) evaluations with the intention to explore new endpoints for targeted therapy
* To find predictive tumour tissue biomarkers for sorafenib/vinflunine treatment
* To evaluate serum and urine markers of apoptosis as potential markers of sorafenib/vinflunine treatment

Rationale/Goal

To evaluate the tolerability and activity of sorafenib combined with vinflunine in patients with advanced or metastatic urothelial cancer.

Tumour biopsies will be collected before and after one cycle of therapy. The translational part of this study aims to explore the predictive value of a number of biomarkers related to the targeted properties of sorafenib and presumptive markers for vinflunine treatment.

In addition, the predictive value of an early functional imaging tracer 18F-FDG-PET/CT will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent;
* histologically confirmed transitional cell (pure or mixed histology including transitional cell carcinoma are allowed) carcinoma of the urothelial tract;
* patients who have received neoadjuvant or adjuvant platinum-containing chemotherapy and who are diagnosed with locoregional recurrent or metastatic disease prior to or at the 6-months" visit , are eligible or
* patients who have received palliative platinum-containing chemotherapy and who are diagnosed with progression prior to or at the 6-months" visit, are eligible or
* patients who have contraindication to platinum-containing chemotherapy;
* previous systemic chemotherapy must have been stopped 14 days before the inclusion with recovery (G1 or less) from any treatment related toxicity;
* measurable and/or non-measurable disease using RECIST and defined as: Measurable disease: lesions that can be measured in at least one dimension and which have not been previously irradiated. Longest diameter 20 mm with conventional techniques or 10 mm with spiral CT scan or MRI. Non-measurable disease: lesions which have not been previously irradiated, or longest diameter <20 mm with conventional techniques or <10 mm with spiral CT scan or MRI, or truly non measurable lesions including bone lesions, ascites, pleural/pericardial effusion, and lymphangitis cutis/pulmonitis;
* age 18 up to 80 years;
* ECOG / WHO Performance Status (PS) ≤1;
* haematological function: haemoglobin ≥100 g/L absolute neutrophil count 1.0 x LL (lower limit of normal value) platelets 100 x 109/L;
* hepatic function: bilirubin <1.5 x ULN*, transaminases <2.5 x ULN*

  *ULN = upper limit of normal value
* renal function: creatinine clearance 40 ml/min (measured by either iohexol clearance or Cr-EDTA technique);
* Clinically normal cardiac function based on ejection fraction (LVEF assessed by MUGA or ECHO, LVEF ≥50%);
* able to swallow and retain oral medication;
* previous treatment related toxicity must be grade ≤1 at time of inclusion and no presence of asthenia, hand-foot skin reaction or rash grade >1 (NCI CTCAE v4.0) at enrolment;
* no known or suspected allergy to the investigational agent or any agents given in association with this trial;

Exclusion Criteria:

* non-transitional cell carcinoma of the urothelial tract (e.g. pure adenocarcinoma or squamous cell carcinoma);
* prior treatment with vinflunine;
* diagnosed brain metastases or leptomeningeal involvement. Brain CT-scans or MRI are not required unless there is clinical suspicion of central nervous system involvement.
* peripheral neuropathy G3 (NCI CTCAE v4.0);
* history of serious or concurrent illness or uncontrolled medical disorder; any medical condition that might be aggravated by treatment or which could not be controlled: active infection requiring antibiotics within 2 weeks before the study inclusion, unstable diabetes mellitus, uncontrolled hypercalcaemia >2.9 mmol/L (or >G2 NCI CTCAE v4.0), concurrent congestive heart failure NYHA (class III-IV) or any type of angina pectoris and/or a diagnosis of myocardial infarction during the previous 6 months and/or poorly controlled hypertension will be excluded, QTc >450 ms at baseline, additional risk factors for Torsade de Pointes (heart failure and hypokalemia (≥G1, i.e. P-K <LLN-2.5 mM) or family history of long QT-syndrome), cardiac arrhythmias requiring anti-arrhythmics (excluding beta-blockers or digoxin for chronic atrial fibrillation);
* patients having received more than one previous systemic chemotherapy for advanced or metastatic disease;
* patients who have received any other investigational or anti-cancer therapy 14 days before the inclusion;
* other malignancies, except adequately treated basal carcinoma of the skin or in-situ cervix carcinoma or incidental prostate cancer (T1a, Gleason score ≤6, PSA <0.5 ng/ml), or any other tumour with a disease free survival of ≥5 years;
* pregnant or lactating women;
* men or women of childbearing potential not employing adequate contraception;
* any psychological, familial, sociological, or geographical condition which does not permit protocol compliance and medical follow-up.
* poorly controlled hypertension. At baseline, blood pressure >150/90 is defined as poorly controlled.
* renal dysfunction: creatinine clearance <40 ml/min measured by either iohexol clearance or Cr-EDTA technique.
* ECOG / WHO Performance Status ≥2
* presence of hand-foot skin reaction or rash >G1 at enrolment;
* known or suspected allergy to the investigational agent or any agents given in association with this trial;
* current medical treatment with any compound that prolongs QTc

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 6 weeks
  Primary endpoint:
  Define the recommended phase II dose (RPTD) by the number of dose limiting toxicity events (recorded during treatment cycle 1 and 2)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Ullén, M.D., Ph.D., Principal Investigator — Dept of Oncology, Karolinska University Hospital
Locations (3):
- Denmark (2):
  - Department of Oncology, Aarhus University Hospital, Aarhus
  - Department of Oncology, Rigshospitalet, Copenhagen
- Department of Oncology, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah CH, Pappot H, Agerbaek M, Holmsten K, Jaderling F, Yachnin J, Gryback P, von der Maase H, Ullen A. Safety and Activity of Sorafenib in Addition to Vinflunine in Post-Platinum Metastatic Urothelial Carcinoma (Vinsor): Phase I Trial. Oncologist. 2019 Jun;24(6):745-e213. doi: 10.1634/theoncologist.2018-0795. Epub 2018 Dec 14. PMID 30552156